CLINICAL TRIAL: NCT03772743
Title: Functional Versus Culprit-only Revascularization in Elderly Patients with Myocardial Infarction and Multivessel Disease
Brief Title: Functional Assessment in Elderly MI Patients with Multivessel Disease
Acronym: FIRE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorzio Futuro in Ricerca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 56/2019/Sper/AOUFe
Record Dates: First submitted 2018-12-09; First posted 2018-12-11 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Myocardial Infarction
Keywords: older adults; multivessel coronary disease; intracoronary physiology; functional assessment
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: All comers, prospective, randomized, multicenter, open-label trial with blinded adjudicated evaluation of outcomes (PROBE).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Culprit-only revascularization (Other): All patients randomized to culprit only revascularization must not undergo percutaneous coronary intervention (PCI) any lesion except from the culprit lesion already treated at the moment of the randomization. Staged procedures are considered protocol violation.
  Interventions: Other: Culprit-only revascularization
- Complete functionally-guided revascularization (Other): Patients who are randomized to this strategy will receive revascularization of the culprit lesion and guided by functional assessment on all non-culprit lesions. Functional evaluation is mandatory for all stenosis with diameter stenosis % between 50 and 90% at visual estimation. Revascularization must be guided by functional assessment on all vessels. The system utilized to obtain functional evaluation is left to Operator's discretion. PCI is allowed only if functional evaluation is positive according to the threshold of the chosen functional system. It is suggested to achieve functional complete revascularization within the index procedure, while it is mandatory to obtain it within the index hospitalization.
  Interventions: Other: Complete functionally-guided revascularization

INTERVENTIONS:
Other: Culprit-only revascularization — Implantation of drug eluting stents with biodegradable polymer with struts ≤65 μ in the culprit lesion of the MI. Each patient should receive revascularization with Supraflex stent or its newer versions
  Arms: Culprit-only revascularization
Other: Complete functionally-guided revascularization — Implantation of drug eluting stents with biodegradable polymer with struts ≤65 μ in the culprit lesion of the MI and in all non culprit lesions with positive functional assessment. Each patient should receive revascularization with Supraflex stent or its newer versions
  Arms: Complete functionally-guided revascularization

SUMMARY:
Elderly patients presenting with myocardial infarction (MI) and multivessel disease are the highest risk population with the worst prognosis. No trial has ever been designed to optimize their outcome. The actual real-life standard of care is, in the best of the cases, culprit only revascularization. However, real-life registries show that outcome of MI elderly patients treated with this strategy is far from being optimal with at least a 15% rate of cardiac death or myocardial infarction at 1 year. To date, studies on this population have been focused on devices (bare metal stent vs biodegradable drug eluting stent) or on dual antiplatelet regimen (long vs short) and no study was focused on evaluating if complete revascularization is able to improve the prognosis in these patients. The contemporary complete revascularization is represented by a functionally-driven revascularization that recently showed to significantly reduce myocardial infarction rate and outperformed an angio-complete revascularization. Thus, our hypothesis is that a functionally-driven complete revascularization in elderly patients with MI and multivessel disease may improve prognosis compared to the actual standard of care in these patients, namely culprit only revascularization. Being a "strategy" trial, we identified the patient-oriented composite endpoint (POCE) as primary outcome of interest (all cause death, any MI, any stroke, any revascularization).

Several pre-specified substudies have been planned. A detailed list of the substudies is available in the website of the trial (http://www.thefiretrial.com)

DETAILED DESCRIPTION:
BACKGROUND OF THE STUDY

Acute myocardial infarction (AMI) is the most frequent clinical presentation in older adults (≥75 years). Registry data shows that up to 65% of patients ≥75 years with AMI has multivessel disease, namely at least one lesion beyond the culprit one with diameter stenosis >50% and located in a coronary artery different from the culprit vessel. Presence of multivessel disease is a marker of worse prognosis. The rate of adverse events, such as death and MI is 3-fold higher in multivessel disease patients if compared to single vessel disease patients. During a 3-5 years follow-up, the number of adverse events related to non-culprit lesions is double than the one related to culprit lesions (data from SWEDEHEART registry and PROSPECT trial). These adverse events are even more frequent in older adults reaching a 15-30% incidence at 1 year. Several studies were focused on older adults with AMI in order to optimize their treatment. The main focus of those studies were: optimal dual antiplatelet therapy (DAPT) duration and type of stent. As for DAPT, data is in favour of a short regimen (1-6 months) as it represents the best balance between ischemic protection and reduction of bleeding events. In both LEADERS FREE and ZEUS trials, age was the main criteria for enrollment and it was considered as a marker of high risk of bleeding event. In the ongoing XIENCE 28 study, age ≥75 years is considered a sufficient criteria to prescribe 28 days of DAPT after stent implantation.

As for stent type, the recent SENIOR trial showed that biodegradable polymer second generation drug eluting stents (DES) are the gold standard in older adults receiving percutaneous coronary interventions (PCI). These stents clearly outperformed bare metal stents with a low event rate in presence of a short DAPT regimen. Thus, at the present time, we have sufficient data to consider biodegradable polymer DES and short DAPT as cornerstones of the treatment in older adults with MI. On the contrary, we have no scientific evidence regarding the best treatment strategy to apply in multivessel disease patients. It is not clear whether to prefer a culprit only strategy or if revascularization of non-culprit lesions is associated to a reduction of adverse events.

Culprit lesion treatment with PCI and stent implantation in MI setting is universally agreed as gold standard since it reduces morbidity and mortality. In the last 10 years, several studies were focused on the treatment of non-culprit lesions. PRAMI, CULPRIT, DANAMI 3 PRIMULTI, COMPARE ACUTE trial tried to assess if a systematic treatment of non-culprit lesions was associated with an improved prognosis if compared to a culprit only strategy. All these studies showed that complete revascularization clearly reduce the risk of repeated revascularizations. However, no study showed a significant impact on death or MI. When pooled in a meta-analysis, we can observe a trend in favour of MI reduction but data cannot be considered as conclusive. In 2019, COMPLETE trial results will be disclosed. In COMPLETE trial, more than 4000 patients were enrolled with consequent power to detect a difference in terms of death and MI. The limits of all the above mentioned studies are that the mean age was around 60 years and that only ST-segment elevated MI (STEMI) patients were included. No study included a relevant portion of patients ≥75 years nor included no-STEMI (NSTEMI) patients. However, a culprit lesion is identifiable in more than 90% of NSTEMI patients and the issue on their management is similar to the one of the STEMI patients. In addiction, in older adults, clinical presentation is as NSTEMI in more than 70% of the cases. Consequently, it is mandatory to generate solid data on the correct treatment strategy in these patients.

In younger adults (<65 years), in concordance with the solid scientific evidences, it is widespread a complete revascularization strategy. In older adults (≥75 years), also guidelines, in absence of clear data, suggest a case-by-case decision and suggest to consider age as one of the determinants of the final decision (Class IIa level of evidence C, ESC NSTEMI guidelines). Both European and American registry data shows clearly that the most frequently applied strategy is the culprit only one, both in STEMI and NSTEMI patients. Also in the LEADERS FREE trial, patients ≥75 years had multivessel disease in 65% of the cases, but in more than 80% of them, treatment was limited to the culprit lesion. In conclusion, the actual gold standard of treatment in older adults with MI and multivessel disease is the culprit-only strategy. The traditional concept of complete revascularization was based on angiography. Operator visually identified the lesions >50% and decided to treat or not each one of them. Contemporary data on fractional flow reserve and instantaneous free-wave ratio demonstrated that an angio-guided strategy is similar to a coin toss in terms of detection of lesions causing ischemia. This leads to unnecessary PCIs or avoided necessary PCIs in more than 50% of the cases. Studies on angio-complete revascularization probably failed to show an MI reduction because of this reason. In addition, long-term follow-up data of lesions functionally deferred shows that the rate of death and MI at 5 years is below 3%. As a consequence, functional revascularization should be considered as contemporary strategy to achieve a real complete revascularization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥75 years AND
2. MI (ST-segment elevation or not ST.segment elevation MI) with indication to invasive management AND
3. Multi-vessel disease defined as at least 1 non-culprit coronary artery lesion at least 2.5 mm in diameter deemed at visual estimation with a diameter stenosis % ranging from 50 to 99% amenable to successful treatment with PCI AND
4. Successful treatment of culprit lesion

Exclusion Criteria:

1. Planned surgical revascularization
2. Non-cardiovascular co-morbidity reducing life expectancy to < 1 year
3. Any factor precluding 1-year follow-up
4. Prior Coronary Artery Bypass Graft (CABG) Surgery
5. Impossibility to identify a clear culprit lesion
6. Non culprit lesion located in the left main

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1445 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2026-10-03 (Estimated)

PRIMARY OUTCOMES:
Patient oriented cardiac events | 1-year
  cumulative occurrence of all-cause death, any MI, any stroke, any revascularization

SECONDARY OUTCOMES:
Patient oriented cardiac events | 3-year
  cumulative occurrence of all-cause death, any MI, any stroke, any revascularization
Patient oriented cardiac events | 5-year
  cumulative occurrence of all-cause death, any MI, any stroke, any revascularization
Device oriented composite endpoint | 1-year
  cumulative occurrence of Cardiovascular Death, MI or non-culprit target vessel revascularization
Device oriented composite endpoint | 3-year
  cumulative occurrence of Cardiovascular Death, MI or non-culprit target vessel revascularization
Device oriented composite endpoint | 5-year
  cumulative occurrence of Cardiovascular Death, MI or non-culprit target vessel revascularization
Cardiovascular Death or MI | 1-year
  cumulative occurrence of Cardiovascular Death or MI
Cardiovascular Death or MI | 3-year
  cumulative occurrence of Cardiovascular Death or MI
Cardiovascular Death or MI | 5-year
  cumulative occurrence of Cardiovascular Death or MI
All-cause death or MI | 1-year
  cumulative occurrence of All-cause Death or MI
All-cause death or MI | 3-year
  cumulative occurrence of All-cause Death or MI
All-cause death or MI | 5-year
  cumulative occurrence of All-cause Death or MI
All-cause death | 1-year
  cumulative occurrence of All-cause Death
All-cause death | 3-year
  cumulative occurrence of All-cause Death
All-cause death | 5-year
  cumulative occurrence of All-cause Death
MI | 1-year
  cumulative occurrence of MI
MI | 3-year
  cumulative occurrence of MI
MI | 5-year
  cumulative occurrence of MI
Any revascularization | 1-year
  cumulative occurrence of revascularization
Any revascularization | 3-year
  cumulative occurrence of revascularization
Any revascularization | 5-year
  cumulative occurrence of revascularization
Ischemic Adverse Events in patients interrupting DAPT | 1-year
  cumulative occurrence of CV death, MI, stroke and revascularization in patients interrupting DAPT
Ischemic Adverse Events in patients disrupting DAPT | 1-year
  cumulative occurrence of CV death, MI, stroke and revascularization in patients disrupting DAPT
Contrast-Induced Acute Kidney Injury | 1 month
  cumulative occurrence of Contrast-Induced Acute Kidney Injury

OTHER OUTCOMES:
Target Lesion Failure | 1-year
  cumulative occurrence of Target Lesion Failure
Target Lesion Failure | 3-year
  cumulative occurrence of Target Lesion Failure
Target Lesion Failure | 5-year
  cumulative occurrence of Target Lesion Failure
Ischemia-driven Revascularization | 1-year
  cumulative occurrence of ischemia-driven revascularization
Ischemia-driven Revascularization | 3-year
  cumulative occurrence of ischemia-driven revascularization
Ischemia-driven Revascularization | 5-year
  cumulative occurrence of ischemia-driven revascularization
EQ-5D scale | 1-year
  quality of life as assessed by EQ-5D scale
EQ-5D scale | 3-year
  quality of life as assessed by EQ-5D scale
EQ-5D scale | 5-year
  quality of life as assessed by EQ-5D scale
Short Physical Performance Battery | 1-year
  Physical Performance as assessed by Short Physical Performance Battery
Short Physical Performance Battery | 3-year
  Physical Performance as assessed by Short Physical Performance Battery
Short Physical Performance Battery | 5-year
  Physical Performance as assessed by Short Physical Performance Battery
Seattle Angina Questionnarie | 1-year
  angina symptoms control as assessed by Seattle Angina Questionnarie
Seattle Angina Questionnarie | 3-year
  angina symptoms control as assessed by Seattle Angina Questionnarie
Seattle Angina Questionnarie | 5-year
  angina symptoms control as assessed by Seattle Angina Questionnarie

CONTACTS AND LOCATIONS:
Locations (37):
- Italy (22):
  - Ospedale Maggiore, Bologna, Bologna
  - AOU Ferrara, Ferrara, Ferrara
  - Maria Cecilia Hospital, Cotignola, Ravenna
  - Ospedale Santa Maria delle Croci, Ravenna, Ravenna
  - Arcispedale Santa Maria Nuova, Reggio Emilia, Reggio Emilia
  - Ospedale Infermi, Rimini, Rimini
  - ASP Agrigento, Agrigento
  - AOU Sant'Anna e San Sebastiano, Caserta
  - Casa di Cura San Michele Maddaloni, Caserta
  - AO Cannizzaro, Catania
  - Ospedale della Misericordia, Grosseto
  - Ospedale Sant.Andrea, La Spezia
  - AOU Gaetano Martino, Messina
  - Ospedale dell'Angelo, Mestre
  - Ospedale Civile di Baggiovara, Modena
  - Ospedale Santa Croce, Moncalieri
  - AOU Giaccone, Palermo
  - AOU Sant'Andrea, Roma
  - Ospedale SS Annunziata, Savigliano
  - Ospedale Umberto I, Syracuse
  - Ospedale di Rivoli, Torino
  - AOU Integrata di Verona, Verona
- Poland (5):
  - Centrum Kardiologii Inwazyjnej, Elektroterapii i Angiologii, Krosno
  - Centrum Kardiologii Inwazyjnej, Elektroterapii i Angiologii, Nowy Sącz
  - Centrum Kardiologii Inwazyjnej Elektroterapii i Angiologii, Oświęcim
  - Centrum Kardiologii Inwazyjnej, Elektroterapii i Angiologii, Pińczów
  - Podkarpackie Centrum Interwencji Sercowo-Naczyniowych, Sanok
- Spain (10):
  - Complejo Hospitalario de La Coruna, A Coruña
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Clinico San Carlos, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario La FE, Valencia
  - Hospital Clinico Universitario, Valladolid
  - Hospital Alvaro Conqueiro de Vigo, Vigo

IPD SHARING:
Plan to Share IPD: Yes
Data will be available after motivated request to the Executive Committee of the study. All requests will be evaluated for acceptance. Positive evaluation by the Executive Committee is mandatory before data release
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the publication of the manuscripts reporting the primary outcome and the prespecified substudies
Access Criteria: Data will be available after motivated request to the Executive Committee of the study. All requests will be evaluated for acceptance. Positive evaluation by the Executive Committee is mandatory before data release
URL: http://thefiretrial.com

REFERENCES:
- [Background] Biscaglia S, Guiducci V, Santarelli A, Amat Santos I, Fernandez-Aviles F, Lanzilotti V, Varbella F, Fileti L, Moreno R, Giannini F, Colaiori I, Menozzi M, Redondo A, Ruozzi M, Gutierrez Ibanes E, Diez Gil JL, Maietti E, Biondi Zoccai G, Escaned J, Tebaldi M, Barbato E, Dudek D, Colombo A, Campo G. Physiology-guided revascularization versus optimal medical therapy of nonculprit lesions in elderly patients with myocardial infarction: Rationale and design of the FIRE trial. Am Heart J. 2020 Nov;229:100-109. doi: 10.1016/j.ahj.2020.08.007. Epub 2020 Aug 18. PMID 32822656
- [Derived] Sarti A, Erriquez A, Dal Passo B, Casella G, Guiducci V, Moreno R, Escaned J, Marchini F, Cocco M, Verardi FM, Clo S, Caglioni S, Farina J, Barbato E, Vadala G, Cavazza C, Capecchi A, Gallo F, Campo G, Biscaglia S. Complete Revascularization in Older Patients With Myocardial Infarction With or Without Complex Nonculprit Lesions. Circ Cardiovasc Interv. 2025 Nov;18(11):e015902. doi: 10.1161/CIRCINTERVENTIONS.125.015902. Epub 2025 Oct 3. PMID 41039960
- [Derived] Biscaglia S, Erriquez A, Guiducci V, Escaned J, Moreno R, Lanzilotti V, Santarelli A, Cerrato E, Sacchetta G, Menozzi A, Amat-Santos I, Diez Gil JL, Ruozzi M, Barbierato M, Fileti L, Picchi A, Pavasini R, Cimaglia P, Colaiori I, Casella G, Menozzi M, Cavazza C, Caretta G, Scarsini R, D'Amico G, Vadala G, Pilato G, Moscarella E, Tebaldi M, Campo G. Physiology-Guided Complete Revascularization in Older Patients With Myocardial Infarction: Three-Year Outcomes of a Randomized Clinical Trial. JAMA Cardiol. 2025 Nov 1;10(11):1130-1137. doi: 10.1001/jamacardio.2025.3099. PMID 40879426
- [Derived] Cocco M, Campo G, Guiducci V, Casella G, Cavazza C, Cerrato E, Sacchetta G, Moreno R, Menozzi A, Amat Santos I, Diez Gil JL, Scarsini R, Picchi A, Vadala G, Pilato G, Colaiori I, Barbierato M, Arioti M, Pavasini R, Lanzilotti V, Menozzi M, Varbella F, Erriquez A, Biscaglia S. Complete vs Culprit-Only Revascularization in Older Patients With Myocardial Infarction With or Without ST-Segment Elevation. J Am Coll Cardiol. 2024 Nov 12;84(20):2014-2022. doi: 10.1016/j.jacc.2024.07.028. Epub 2024 Aug 31. PMID 39217557
- [Derived] Campo G, Guiducci V, Escaned J, Moreno R, Casella G, Cavazza C, Cerrato E, Contarini M, Arena M, Iniguez Romo A, Gutierrez Ibanes E, Scarsini R, Vadala G, Ando G, Pilato G, Musto d'Amore S, Capecchi A, Trillo Nouche R, Moscarella E, Gambino A, Pavani M, Zanetti A, Pesenti N, Dudek D, Barbato E, Tebaldi M, Biscaglia S. Health-Status Outcomes in Older Patients With Myocardial Infarction: Physiology-Guided Complete Revascularization Versus Culprit-Only Strategy. Circ Cardiovasc Qual Outcomes. 2024 Jul;17(7):e010490. doi: 10.1161/CIRCOUTCOMES.123.010490. Epub 2024 Jun 18. PMID 38887951
- [Derived] Erriquez A, Campo G, Guiducci V, Casella G, Menozzi M, Cerrato E, Sacchetta G, Moreno R, Arena M, Amat Santos I, Diez Gil JL, Scarsini R, Ruozzi M, Arioti M, Picchi A, Barbierato M, Moscarella E, Musto D'Amore S, Lanzilotti V, Cavazza C, Rezzaghi M, Cocco M, Marrone A, Verardi FM, Escaned J, Barbato E, Colaiori I, Pesenti N, Carrara G, Biscaglia S. QFR for the Revascularization of Nonculprit Vessels in MI Patients: Insights From the FIRE Trial. JACC Cardiovasc Interv. 2024 Jun 24;17(12):1425-1436. doi: 10.1016/j.jcin.2024.04.022. Epub 2024 May 14. PMID 38752972
- [Derived] Erriquez A, Campo G, Guiducci V, Escaned J, Moreno R, Casella G, Menozzi M, Cerrato E, Sacchetta G, Menozzi A, Santos IA, Ibanes EG, Scarsini R, Vadala G, Ando G, Diez-Gil JL, d'Amore SM, Capecchi A, Colaiori I, Gallo F, Pavasini R, Marrone A, Pompei G, Lanzilotti V, Dudek D, Barbato E, Tebaldi M, Biscaglia S. Complete vs Culprit-Only Revascularization in Older Patients With Myocardial Infarction and High Bleeding Risk: A Randomized Clinical Trial. JAMA Cardiol. 2024 Jun 1;9(6):565-573. doi: 10.1001/jamacardio.2024.0804. PMID 38717753
- [Derived] Pavasini R, Campo G, Serenelli M, Tonet E, Guiducci V, Escaned J, Moreno R, Casella G, Cavazza C, Varbella F, Sacchetta G, Arena M, Santos IA, Ibanes EG, Scarsini R, D'Amico G, Ruiz-Poveda FL, Diez Gil JL, Pignatelli G, Iannopollo G, Colaiori I, Santos RC, Marrone A, Fileti L, Rigattieri S, Barbato E, Ocaranza-Sanchez R, Biscaglia S. Impact of pre-admission physical activity on benefits of physiology-guided complete revascularization in older patients with myocardial infarction: insights from the FIRE trial. Eur J Prev Cardiol. 2024 Sep 6;31(12):1451-1459. doi: 10.1093/eurjpc/zwae069. PMID 38452238
- [Derived] Biscaglia S, Guiducci V, Escaned J, Moreno R, Lanzilotti V, Santarelli A, Cerrato E, Sacchetta G, Jurado-Roman A, Menozzi A, Amat Santos I, Diez Gil JL, Ruozzi M, Barbierato M, Fileti L, Picchi A, Lodolini V, Biondi-Zoccai G, Maietti E, Pavasini R, Cimaglia P, Tumscitz C, Erriquez A, Penzo C, Colaiori I, Pignatelli G, Casella G, Iannopollo G, Menozzi M, Varbella F, Caretta G, Dudek D, Barbato E, Tebaldi M, Campo G; FIRE Trial Investigators. Complete or Culprit-Only PCI in Older Patients with Myocardial Infarction. N Engl J Med. 2023 Sep 7;389(10):889-898. doi: 10.1056/NEJMoa2300468. Epub 2023 Aug 26. PMID 37634150